CLINICAL TRIAL: NCT02100969
Title: Open Label Study of Subcutaneous Immunoglobulin (SCIg) in Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mazen Dimachkie, MD (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, Mazen Dimachkie, MD, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001041
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Myasthenia Gravis
Keywords: MG; Hizentra; autoimmune neuromuscular disorder
MeSH Terms: conditions — Myasthenia Gravis | interventions — Hizentra; gamma-Globulins; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIZENTRA ® (Experimental): Hizentra is a subcutaneous (under the skin) immunoglobin (SCIg). Participants will receive Hizentra in a minimum of one infusion per week and a maximum of 4 infusions per week. Dose and rate depend on the visit and how each participant tolerates the drug. Max cc per site is 50 cc per site per hour.
  Interventions: Drug: HIZENTRA ®

INTERVENTIONS:
Drug: HIZENTRA ® — Patients must fulfill inclusion criteria and remain stable at week 0, which means QMG does not increase by 3 points, will enter receive Hizentra for 12 weeks.
  Other Names: Immune Globulin Subcutaneous (Human), 20% Liquid

SUMMARY:
The purpose of this study is to determine whether Hizentra is a safe and effective treatment for people with myasthenia gravis (MG).

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is a rare autoimmune disorder which causes the muscles to become weak because the immune system attacks the connection between the nerves and the muscles.

Hizentra is a subcutaneous (under the skin) immunoglobin (SCIg). An immunoglobin is a blood protein. Hizentra is being studied for the treatment of patients with MG. Hizentra is administered by an injection into the skin through a portable infusion pump, which may be easier for patients to administer than the current treatments.

Participants will be asked to complete 9 clinic visits and 3 telephone calls. It could take up to 30 weeks to complete all study visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 and older
* Patients must have prior or current documentation of MGFA MG grades 2, 3, or 4 generalized MG, according to the MGFA classification system.48 These grades correspond to mild (2), moderate (3), and severe (4)
* Elevated AChR or MuSK Ab. These tests will have been performed at some time prior to entry into the study. Double seronegative MG patients with prior documentation of an abnormal decrement (>10%) on slow repetitive nerve stimulation or an abnormal single fiber EMG will also be allowed to participate
* Patient's signs and symptoms should not be better explained by another disease process.
* IVIg maintenance dose of 0.2 to 2 gm/kg/4 weeks or equivalent dose administered Q 2-4 weeks±3days
* Stable IVIg for at least 3 cycles (definition of stability: no change in prescribed dosage or frequency by the treating physician)
* Patient must be receiving no more than 200g/4weeks of IVIg.
* Patients must be willing to complete the study and return for follow-up visits.
* Patients must be willing to give written informed consent before participating in this study. A copy of the signed consent must be kept in the patient's medical record.
* Patients can be on the following drugs as long as there has been no dose change for 60 days: azathioprine, cyclosporine, cyclophosphamide, mycophenolate mofetil, tacrolimus, methotrexate or other immunosuppressive drugs.
* Patients can be on prednisone as long as there has been no dose change for 30 days.

Exclusion Criteria:

* MGFA grade V within 6 months of screening.
* A history of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue.
* Other major chronic or debilitating illnesses within six months prior to study entry.
* Female patients who are premenopausal and are: (a) pregnant on the basis of a serum pregnancy test, (b) breast-feeding, or (c) not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures).
* Altered levels of consciousness, dementia, or abnormal mental status.
* Thymectomy in the previous three months.
* Evidence of renal insufficiency (Cr>1.5 x elevated) or liver disease (transaminases > 2.5 x elevation) at screening.
* Skin disease that would interfere with assessment of injection site reaction
* History of severe reactions to IVIg or SCIg.
* Participation in a research study within the last 3 months
* Treatment with rituximab or other biologics within 12 months of study entry
* Inability to provide informed consent.
* History of thrombotic episodes within the last year prior to enrollment
* Known allergic or other severe reactions to blood products including intolerability to previous normal human immunoglobulin for intravenous administration (IVIG) and/or subcutaneous immunoglobulin (SCIG), such as history of clinically relevant hemolysis after IVIG infusion, aseptic meningitis, recurrent severe headache, hypersensitivity, severe generalized or severe local skin reaction.
* History of IgA deficiency or evidence of IgA deficiency at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen M Dimachkie, MD, Principal Investigator — University of Kansas Medical Center
Locations (5):
- United States (4):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of Kansas Medical Center, Kansas City, Kansas
  - University at Buffalo, Buffalo, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- University of Toronto, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: North American study involving 5 sites (4 in the US and 1 in Canada). Subjects were recruited through clinical practice and advertisement through the Myasthenia Gravis Foundation of America.
Groups:
- Privigen/Hizentra: Privigen: 3 rounds of IV privigen was infused every 4 weeks until baseline visit week 0.
  Hizentra: Hizentra infused sub cutaneously based on weight and subject prescribed dose.
Period: Overall Study
Arm/Group | Privigen/Hizentra
Started | 23
Completed | 22
Not Completed | 1
Not completed — Did not pass screening phase | 1

BASELINE CHARACTERISTICS:
Groups:
- Hizentra: Hizentra is a subcutaneous (under the skin) immunoglobin (SCIg). Participants will receive weekly Hizentra. Dose and rate depend on the visit and how each participant tolerates the drug. Max flow rate not to exceed 100 mL per hour.
  HIZENTRA ®
Arm/Group | Hizentra
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.36 (17.001)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 18
  Race: African American | 2
  Race: Asian | 1
  Race: Other | 1
  Race: Unknown | 1
Region of Enrollment [Number; unit: participants]
  Canada | 11
  United States | 12
Quantitative Myasthenia Gravis test at Baseline [Median (Inter-Quartile Range); unit: points] — The QMG is a clinical composite scale administered by a physician or trained clinical evaluator. The QMG scores 13 different assessments that align with common symptoms of MG. Each item is graded on a scale of 0 - 3. The QMG has a total score of 0 - 39 with 0 being the best (no symptoms) and 39 being the worst (severe symptoms). Population: As per the protocol, only those patients who completed the screening phase are eligible for analysis. In our case this is 22 out of 23 patients.
  points
    number analyzed (Participants) | 22
    (all) | 10 [6.75 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Whose Quantitative Myasthenia Gravis Scores Are Increased by no More Than 3 Points at the End of the SCIg Treatment Phase
Description: The QMG is a 13 item ordinal scale which measures ocular, bulbar, extremity fatigue and strength, along with respiratory function. The scale is from 0 - 3 for each item, with 0 meaning normal and 3 is severe. Total score can range from 0 to 39.
  Change in MG severity will be measured using the Quantitative Myasthenia Gravis (QMG) Score for Disease severity. The QMG is a validated clinical composite scale. As mentioned in the protocol, our hypotheses are:
  H0: Proportion of patients whose QMG scores are increased by more than 3 points at the end of the SCIg treatment phase ≤ 0.65 HA: Proportion of patients whose QMG scores are increased by no more than 3 points at the end of the SCIg treatment phase > 0.65
  Thus, analysis of the primary outcome is done as a one-sample Z test of proportions. That is, the QMG is a continuous outcome, but analyses results are reported as proportions.
Time Frame: Change from Baseline to Week 12
Population: 23 patients were enrolled in the study. The protocol mentions that only those subjects who have stable QMG in the screening phase will be considered eligible for analyses. In our case 22 out of 23 patients are eligible for the final analyses.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Hizentra
Number analyzed (Participants) | 22
proportion of participants | 0.864 [0.720 to 1.000]
Statistical Analysis 1: Comparison: Hizentra; Sample size/power calculations are mentioned in the study protocol. The study hypotheses are as follows: H0: Proportion of patients whose QMG scores are increased by no more than 3 points at the end of the SCIg treatment phase ≤ 0.65 HA: Proportion of patients whose QMG scores are increased by no more than 3 points at the end of the SCIg treatment phase > 0.65; Test type: Superiority; p = 0.0179, One sample Z test of proportions — No adjustment is required as we are not doing multiple comparisons for the primary outcome analyses; proportion of "successes" = 0.864, 95% CI 2-sided [0.720 to 1.000] — One sample Z test of proportions is used. Method of handling missing data (as per protocol) is Last Observation Carried Forward (LOCF). Only 2 participants had missing values and in our case the LOCF results reflect a 'best-case' scenario

2. Secondary Outcome: Myasthenia Gravis-specific Activities of Daily Living Scale (MG-ADL) Scores
Description: Myasthenia Gravis-specific Activities of Daily Living scale (MG-ADL): Composite measure of scores from measurement scales. The MG-ADL has a scale of 0 - 24 with 0 being the lowest (no symptoms) and 24 being the highest (most severe symptoms. The MG-ADL is a staff-administered, patient-reported questionnaire that measures 8 commons symptoms of myasthenia gravis and grades them on a scale of 0 - 3.
Time Frame: Change from Baseline to Week 12
Population: Here we consider the 22 participants on whom the MG-ADL scores at either baseline or Week 12 are available for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 22
score on a scale
  Week 12: number analyzed (Participants) | 20
  Week 12 | 3 [0 to 4.5]
  Baseline | 3 [1 to 7]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.113, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 0 — The value of the signed rank test statistic is 44.50

3. Secondary Outcome: Myasthenia Gravis Quality of Life (MG QOL-15) Scores
Description: MG Quality of Life (QOL)-15: Composite measure of scores from measurement scales. The MG QOL-15 is a questionnaire answered by the patient that asked about different symptoms of MG. The questionnaire consists of 15 questions that are graded on a scale of 0 - 4. The total score has a range of 0 - 60 with a higher score meaning more severe symptoms or a worse outcome.
Time Frame: Change from Baseline to Week 12
Population: Here we consider the 22 participants on whom the MG-ADL scores at either baseline or Week 12 are available for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 22
score on a scale
  Week 12: number analyzed (Participants) | 20
  Week 12 | 16 [6.5 to 32.75]
  Baseline | 22 [9 to 28.50]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.612, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 6

4. Secondary Outcome: Myasthenia Gravis Composite (MGC) Score
Description: The MGC takes scores from the MG-ADL, the QMG, and combines them will manual muscle testing scores to create the MGC. The scale of this score ranges from 0 - 50 with higher scores meaning a worse outcome or more sever symptoms.
Time Frame: Change from Baseline to Week 12
Population: Here we consider the 21 participants on whom the MG-Composite scores are available for analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 21
score on a scale
  Week 12: number analyzed (Participants) | 20
  Week 12 | 4 [0.25 to 10.75]
  Baseline | 6 [1 to 12]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.047, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 2 — The value of the signed-rank test statistic is 53

5. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - Convenience Score
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) - Convenience Score measured on a scale of 0 to 100. 0 indicates no treatment convenience satisfaction and 100 indicates highest treatment convenience satisfaction.
Time Frame: Change from Baseline to Week 12
Population: This secondary outcome was recorded for 18 patients. Analysis is done as per the protocol.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 18
score on a scale
  Week 12 | 75 [47.20 to 81.90]
  Baseline | 69.40 [51.40 to 77.80]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.901, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 5.60

6. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - Effectiveness Score
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) - Effectiveness Score measured on a scale of 0 to 100. 0 indicates no treatment effectiveness satisfaction and 100 indicates highest treatment effectiveness satisfaction.
Time Frame: Change from Baseline to Week 12
Population: This secondary outcome was recorded for 20 patients. Analysis is done as per the protocol.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 20
score on a scale
  Week 12 | 79.20 [52.10 to 100]
  Baseline | 75 [50 to 83.30]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.510, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 4.20

7. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - Satisfaction Score
Description: Treatment Satisfaction Questionnaire for Medication (TSQM) - Satisfaction Score measured on a scale of 0 to 100. 0 indicates no treatment satisfaction and 100 indicates highest treatment satisfaction.
Time Frame: Change from Baseline to Week 12
Population: This secondary outcome was recorded for 18 patients. Analysis is done as per the protocol.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Hizentra
Number analyzed (Participants) | 18
score on a scale
  Week 12 | 83.30 [45.80 to 91.70]
  Baseline | 75 [58.30 to 97.90]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.289, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 8.30

8. Secondary Outcome: Immunoglobulin G (IgG) Antibody Levels
Description: Measure IgG level (mg/dL) between intravenous and subcutaneous study phases. Normal range equals 762-1488 mg/dL.
Time Frame: Change from "Week -10 to Week 0" versus "Week 1 to Week 12"
Population: Note: Change in IgG from Week -10 to Week 0 can be assessed for 20 participants. Change in IgG from Week 1 to Week 12 can be assessed for 19 participants.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Hizentra
Number analyzed (Participants) | 20
mg/dL
  Change: Week -10 to Week 0 | 661 [496.25 to 981]
  Change: Week 1 to Week 12: number analyzed (Participants) | 19
  Change: Week 1 to Week 12 | -54 [-423 to 150]
Statistical Analysis 1: Comparison: Hizentra; Test type: Superiority; p = 0.0028, Wilcoxon Signed Rank for paired data; Median Difference (Net) = 715

9. Secondary Outcome: Tolerabililty
Description: Tolerability is assessed as the number of subjects who completed the study and/or did not withdraw due to worsening.
Time Frame: 12 weeks from start of SCIg
Measure: Count of Participants; unit: Participants
Arm/Group | HIZENTRA ®
Number analyzed (Participants) | 22
Participants | 20

ADVERSE EVENTS:
Time Frame: 23 weeks
Groups:
- Privigen/Hizentra: Experimental Treatment arm: Privigen/Hizentra assigned to subjects who are stable in the screening phase of the study.
Arm/Group | Privigen/Hizentra
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Privigen/Hizentra (N=23)
Thromboembolic event (Vascular disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
Psychiatric Disorders- Other (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Privigen/Hizentra (N=23)
Injection Site Reactions (Skin and subcutaneous tissue disorders) | 3 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3)
Headache (Nervous system disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Blood and Lymphatic System Disorder (Blood and lymphatic system disorders) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Neck edema (General disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial Infection (Infections and infestations) | 1 (1)
Edema Limbs (General disorders) | 1 (4)
Eye Disorders (Eye disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1)
Pain Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Musculoskeletal and Connective Tissue Disorder Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 1 (1) — Increased Creatinine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02100969/Prot_001.pdf
  • Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02100969/SAP_000.pdf